## Cover Letter:

All enclosed below documents are part of the clinical trial NCT03536819

Study Name: Radio-frequency rejuvenation for pelvic floor and vagina

Protocol No.: DO607404A

Document date: September 20, 2017

**SPONSOR**: InMode Ltd.

Tabor House

Industrial Park South

Yokneam 20692 ISRAEL

POB 44

Tel +972-4-9097309

Fax +972-4-9096310

## I. Data analysis.

## A. Analysis Sets

- 1. Safety Analysis Set
  - a) The safety analysis set will include all subjects using Votiva procedures at least a single time.
- 2. Performance Analysis Set
  - a) Performance analysis set will consist of all subjects providing at least one post treatment performance measurement.
- 3. Treatment of Missing Values
  - a) Only observed data will be used; i.e. missing data will not be imputed.

## B. Statistical Analysis

 Means, and standard deviations for each characteristic will be calculated. Paired sample t-test will be computed to assess changes in before treatment and follow-up scores. Statistical significance will be calculated and two-tail significance level of 0.05 will be used. All analyses will be conducted using IBM SPSS 21.0.